CLINICAL TRIAL: NCT02337751
Title: A Multicenter, Open-label, Long-term, Extension, Phase 3 Study to Evaluate the Safety and Efficacy of TVP-1012 at 1 mg in Early Parkinson's Disease Patients Not Treated With Levodopa
Brief Title: A Phase 3, Long-term, Extension Study of TVP-1012 (1 mg) in Early Parkinson's Disease Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TVP-1012/OCT-001; U1111-1165-1437 (Registry Identifier: WHO); JapicCTI-152761 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TVP-1012 1mg Group (Experimental): TVP-1012 (1 mg/day) once daily, either before or after breakfast.
  Interventions: Drug: TVP-1012 1mg

INTERVENTIONS:
Drug: TVP-1012 1mg — TVP-1012 1mg Tablets

SUMMARY:
The purpose of this study is to evaluate the long-term safety of TVP-1012 (1 mg/day) in Japanese participants with early Parkinson's disease.

DETAILED DESCRIPTION:
This is a multicenter, open-label, long-term, extension, phase 3 study to evaluate the safety and efficacy of long-term administration of TVP-1012 at 1 mg for another 26 weeks in participants with early Parkinson's disease who have completed the preceding TVP-1012/CCT-001 (NCT02337725) study.

Among participants of the TVP-1012/CCT-001 study, those consenting to participate in this study prior to complete the preceding study and fulfilling the eligibility criteria will be enrolled in this study. From the day after the Visit 8 of the preceding study, participants will receive 1 mg of TVP-1012 once daily for 26 weeks in an unblinded manner.

ELIGIBILITY:
Inclusion Criteria:

* The participant has completed the preceding study.
* The participant has shown no safety issues during the study treatment in the preceding study, in the opinion of the investigator or subinvestigator.

Exclusion Criteria:

* The participant has undergone blood collection of >= 400 mL within 90 days prior to the start of treatment in this study.
* The participant is required to take any of the excluded medications or treatments.
* The participant is required surgery or hospitalization for surgery during the study period.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (56):
- Japan (56):
  - Nagoya, Aichi-ken
  - Matsuyama, Ehime
  - Tōon, Ehime
  - Kitakyushu, Fukuoka
  - Ōnojō, Fukuoka
  - Asahikawa, Hokkaido
  - Iwamizawa, Hokkaido
  - Akashi, Hyōgo
  - Kobe, Hyōgo
  - Tsuchiura, Ibaraki
  - Tsukuba, Ibaraki
  - Ichinoseki, Iwate
  - Morioka, Iwate
  - Takamatsu, Kagawa-ken
  - Fujisawa, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Gōshi, Kumamoto
  - Sendai, Miyagi
  - Matsumoto, Nagano
  - Nishisonogi, Nagasaki
  - Sonogishukugō, Nagasaki
  - Tenri, Nara
  - Jōetsu, Niigata
  - Higashiosaka, Osaka
  - Suita, Osaka
  - Takatsuki, Osaka
  - Toyonaka, Osaka
  - Irima, Saitama
  - Fuji, Shizuoka
  - Hamamatsu, Shizuoka
  - Izunokuni, Shizuoka
  - Shimono, Tochigi
  - Yoshinogawa, Tokushima
  - Bunkyo-ku, Tokyo
  - Fuchū, Tokyo
  - Kodaira, Tokyo
  - Meguro-ku, Tokyo
  - Nerima-ku, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Akita
  - Aomori
  - Fukuoka
  - Fukushima
  - Hiroshima
  - Kochi
  - Kyoto
  - Niigata
  - Okayama
  - Osaka
  - Tokushima
  - Toyama
  - Wakayama
  - Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Hattori N, Takeda A, Takeda S, Nishimura A, Kitagawa T, Mochizuki H, Nagai M, Takahashi R. Long-term, open-label, phase 3 study of rasagiline in Japanese patients with early Parkinson's disease. J Neural Transm (Vienna). 2019 Mar;126(3):299-308. doi: 10.1007/s00702-018-1964-3. Epub 2019 Jan 28. PMID 30689042

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 68 investigative sites in Japan, from 10 July 2015 to 14 March 2017.
Pre-assignment Details: All participants with Parkinson's disease who completed the 26-week treatment period in preceding study (TVP-1012/CCT-001: NCT02337725) were enrolled in this study. Participants in TVP-1012 group and in Placebo group in preceding study were assigned to TVP-1012+TVP-1012 Group and Placebo+TVP-1012 Group in this study, respectively.
Groups:
- Placebo + TVP-1012 Group: TVP-1012 (1 mg/day) once daily, either before or after breakfast for up to 26 weeks. Reported data on Participants Flow was all participants who enrolled in this study and had assigned to Placebo group in preceding study.
- TVP-1012 + TVP-1012 Group: TVP-1012 (1 mg/day) once daily, either before or after breakfast for up to 26 weeks. Reported data on Participants Flow was all participants who enrolled in this study and had assigned to TVP-1012 group in preceding study.
Period: Overall Study
Arm/Group | Placebo + TVP-1012 Group | TVP-1012 + TVP-1012 Group
Started | 95 | 103
Completed | 84 | 87
Not Completed | 11 | 16
Not completed — Pretreatment Event/Adverse Event | 2 | 3
Not completed — Voluntary Withdrawal | 6 | 8
Not completed — Lack of Efficacy | 2 | 5
Not completed — Investigator's Judgement | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set; All participants who received at least one dose of TVP-1012 during this study and/or the preceding study (TVP-1012/CCT-001: NCT02337725). The analysis set included 103 participants who enrolled in this study and 14 participants who enrolled only in TVP-1012/CCT-001 and received TVP-1012 (totally 117 participants).
Groups:
- Placebo + TVP-1012 Group: Placebo, once daily, either before or after breakfast in preceding study for 26 weeks, followed by in this study, TVP-1012 (1 mg/day) once daily, either before or after breakfast for 26 weeks.
- TVP-1012 + TVP-1012 Group: TVP-1012 1 mg, once daily, either before or after breakfast in preceding study for 26 weeks, followed by in this study, TVP-1012 (1 mg/day) once daily, either before or after breakfast for 26 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo + TVP-1012 Group | TVP-1012 + TVP-1012 Group | Total
Number analyzed (Participants) | 95 | 117 | 212
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (9.13) | 67.4 (8.99) | 66.5 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 64 | 117
  Male | 42 | 53 | 95
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 95 | 117 | 212
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 159.2 (9.28) | 158.9 (8.87) | 159.0 (9.04)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 56.68 (9.773) | 57.91 (11.803) | 57.36 (10.932)
BMI [Mean (Standard Deviation); unit: kg/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/meter (m)^2 | 22.28 (2.798) | 22.78 (3.303) | 22.56 (3.090)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 56 | 63 | 119
  Current Smoker | 7 | 5 | 12
  Ex-Smoker | 32 | 49 | 81
Timing of Study Drug Dose [Count of Participants; unit: Participants]
  Before Breakfast | 48 | 59 | 107
  After Breakfast | 47 | 58 | 105
Duration of Parkinson's Disease [Mean (Standard Deviation); unit: Years] | 1.52 (1.223) | 1.97 (1.981) | 1.77 (1.695)
Modified Hoehn & Yahr Stage [Mean (Standard Deviation); unit: Units on a scale] — Modified Hoehn & Yahr Stage represented severity for symptoms of Parkinson's disease progress. The Stage of Modified Hoehn & Yahr were assigned from Stage 0 (Asymptomatic) to Stage 5 (Wheelchair bound or bedridden unless aided (unable to walk even if aided)).
  Units on a scale | 2.13 (0.627) | 2.18 (0.628) | 2.16 (0.627)
MDS-UPDRS Part II + Part III Total Score (Pre-Dose) [Mean (Standard Deviation); unit: Scores on a scale] — Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) retained the four-scale structure with a reorganization of the various subscales: (Part I) non-motor experiences of daily living (13 items), (Part II) motor experiences of daily living (13 items), (Part III) motor examination (18 items), and (Part IV) motor complications (6 items). Each subscale had 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range for Part II+III Total Score was 0-188, with the higher score reflecting the greater severity.
  Scores on a scale | 33.0 (15.86) | 34.4 (16.95) | 33.8 (16.44)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Description: Reported data was the number collected from the first dose of TVP-1012 to the end of study (up to 52 weeks). Timeframe was 52 weeks that was total duration of both this study (26 weeks) and the preceding study (TVP-1012/CCT-001: NCT02337725; 26 weeks).
Time Frame: Up to 52 weeks
Population: Safety Analysis Set: All participants who received at least 1 dose of TVP-1012 during this study and/or the preceding study (TVP-1012/CCT-001: NCT02337725). The analysis set included 103 participants who enrolled in this study and 14 participants who enrolled only in TVP-1012/CCT-001 and received TVP-1012 (totally 117 participants).
Measure: Count of Participants; unit: Participants
Groups:
- Placebo + TVP-1012 Group: Placebo, once daily, either before or after breakfast in preceding study for 26 weeks, followed by in this study, TVP-1012 (1 mg/day) once daily, either before or after breakfast for up to 26 weeks.
- TVP-1012 + TVP-1012 Group: TVP-1012 1 mg, once daily, either before or after breakfast in preceding study for 26 weeks, followed by in this study, TVP-1012 (1 mg/day) once daily, either before or after breakfast for up to 26 weeks.
Arm/Group | Placebo + TVP-1012 Group | TVP-1012 + TVP-1012 Group
Number analyzed (Participants) | 95 | 117
Participants | 51 | 91

2. Secondary Outcome: Number of Participants With TEAE Related to Clinical Laboratory Tests
Description: as for outcome 1
Time Frame: Up to 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + TVP-1012 Group | TVP-1012 + TVP-1012 Group
Number analyzed (Participants) | 95 | 117
Participants
  Blood Creatine Phosphokinase Increased | 0 | 1
  Blood Triglycerides Increased | 1 | 0
  Blood Urine Present | 1 | 0
  C-Reactive Protein Increased | 0 | 1
  Glycosylated Haemoglobin Increased | 0 | 1
  Liver Function Test Abnormal | 0 | 1
  Liver Function Test Increased | 0 | 1
  White Blood Cell Count Increased | 1 | 0

3. Secondary Outcome: Number of Participants With Markedly Abnormal Vital Signs Values
Description: Reported data was the number collected from the first dose of TVP-1012 to the end of study (up to 52 weeks). Here "mmHg" is Millimeter of mercury. Timeframe was 52 weeks that was total duration of both this study (26 weeks) and the preceding study (TVP-1012/CCT-001: NCT02337725; 26 weeks).
Time Frame: Up to 52 weeks
Population: Safety Analysis Set: All participants who received at least 1 dose of TVP-1012 during this study, 103 participants, and only in the preceding study (TVP-1012/CCT-001: NCT02337725), 14 participants, totally 117 participants.
  The number of participants analyzed for each items are participants evaluable for each item within the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + TVP-1012 Group | TVP-1012 + TVP-1012 Group
Number analyzed (Participants) | 95 | 117
Participants
  Temperature <35.6 Celsius (ºC): number analyzed (Participants) | 95 | 116
  Temperature <35.6 Celsius (ºC) | 13 | 30
  Temperature >37.7 ºC: number analyzed (Participants) | 95 | 116
  Temperature >37.7 ºC | 0 | 1
  Systolic Blood Pressure <90 mmHg: number analyzed (Participants) | 95 | 116
  Systolic Blood Pressure <90 mmHg | 3 | 3
  Diastolic Blood Pressure <50 mmHg: number analyzed (Participants) | 95 | 116
  Diastolic Blood Pressure <50 mmHg | 4 | 0
  Diastolic Blood Pressure >100 mmHg: number analyzed (Participants) | 95 | 116
  Diastolic Blood Pressure >100 mmHg | 6 | 13
  Pulse <45 Beats per Minute (bpm): number analyzed (Participants) | 95 | 116
  Pulse <45 Beats per Minute (bpm) | 0 | 1

4. Secondary Outcome: Number of Participants With TEAE Related to Electrocardiograms (ECG) (ECG QT Prolonged)
Description: as for outcome 1
Time Frame: Up to 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + TVP-1012 Group | TVP-1012 + TVP-1012 Group
Number analyzed (Participants) | 95 | 117
Participants | 1 | 1

5. Secondary Outcome: Number of Participants With TEAE Related to Body Weight (Weight Loss)
Description: as for outcome 1
Time Frame: Up to 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + TVP-1012 Group | TVP-1012 + TVP-1012 Group
Number analyzed (Participants) | 95 | 117
Participants | 1 | 0

6. Secondary Outcome: Change From Baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II + Part III Total Score
Description: MDS-UPDRS retains the four-scale structure with a reorganization of the various subscales. The scales are now titled; (Part I) non-motor experiences of daily living (13 items), (Part II) motor experiences of daily living (13 items), (Part III) motor examination (18 items), and (Part IV) motor complications (six items). Each subscale now has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range for Part II+III Total Score was 0-188, with the higher score reflecting the greater severity. Timeframe was 52 weeks that was total duration of both this study (26 weeks) and the preceding study (TVP-1012/CCT-001: NCT02337725; 26 weeks).
Time Frame: Baseline to End of treatment (Week 52)
Population: Full Analysis Set (FAS); All randomized participants who received at least one dose of TVP-1012 during this study, 103 participants, and only in the preceding study (TVP-1012/CCT-001: NCT02337725), 14 participants, totally 117 participants. The analyzed numbers for each arm were participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- TVP-1012 +TVP-1012 Group: TVP-1012 1 mg, once daily, either before or after breakfast in preceding study for 26 weeks, followed by in this study, TVP-1012 (1 mg/day) once daily, either before or after breakfast for up to 26 weeks.
Arm/Group | Placebo + TVP-1012 Group | TVP-1012 +TVP-1012 Group
Number analyzed (Participants) | 95 | 117
Units on a Scale | -2.8 (6.01) | -2.8 (9.62)

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: At each visit investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by participant or observed by investigator was recorded, irrespective of the relation to study treatment. On adverse events table, only events that occurred after at least one dose of TVP-1012 during this study, 103 participants, and only in the preceding study (TVP-1012/CCT-001: NCT02337725), 14 participants, totally 117 participants, were reported.
Arm/Group | Placebo + TVP-1012 Group | TVP-1012 + TVP-1012 Group
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/117
Serious Adverse Events (participants affected / at risk) | 4/95 | 6/117
Other Adverse Events (participants affected / at risk) | 23/95 | 49/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + TVP-1012 Group (N=95) | TVP-1012 + TVP-1012 Group (N=117)
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Leukoplakia oral (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Microscopic polyangiitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + TVP-1012 Group (N=95) | TVP-1012 + TVP-1012 Group (N=117)
Nasopharyngitis (Infections and infestations) | 17 | 31
Fall (Injury, poisoning and procedural complications) | 6 | 11
Contusion (Injury, poisoning and procedural complications) | 5 | 5
Headache (Nervous system disorders) | 1 | 7
Eczema (Skin and subcutaneous tissue disorders) | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT02337751/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT02337751/SAP_001.pdf